CLINICAL TRIAL: NCT02255721
Title: Healthy Sleep Intervention For Preschool Children: A Randomized Controlled Trial of the SHIP Intervention
Brief Title: Sleep Health in Preschoolers: a Randomized Controlled Trial
Acronym: SHIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michelle Garrison, Research Assistant Professor, University of Washington, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 416530030101; R01HD071937 (NIH)
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Ships

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SHIP Intervention (Experimental): SHIP is a health behavior change intervention to give parents the knowledge, motivation, and skills necessary to set goals, problem-solve, and improve their child's sleep.
  Interventions: Behavioral: SHIP (Sleep Health in Preschoolers)
- SHIP Control Arm (Active Comparator): The active control arm uses the same strategies as the SHIP intervention arm, but for child health topics unrelated to sleep or outcome measures.
  Interventions: Behavioral: SHIP Control Arm

INTERVENTIONS:
Behavioral: SHIP (Sleep Health in Preschoolers) — SHIP (Sleep Health in Preschoolers) is a family-centered health behavior change intervention for child behavioral sleep problems delivered 1:1 to parents via a home visit and follow-up phone calls.
  Arms: SHIP Intervention
Behavioral: SHIP Control Arm — Families will receive a family-centered health behavior change intervention for child health topics unrelated to sleep or outcome measures, delivered 1:1 to parents via a home visit and follow-up phone calls.
  Arms: SHIP Control Arm

SUMMARY:
The SHIP study is a randomized controlled trial of an intervention for preschool children with sleep problems, in which we aim to give parents the knowledge, motivation, and skills necessary to set goals, problem-solve, and improve their child's sleep. In collecting three years of follow-up data, we will be able to determine the impact of the SHIP intervention on childhood sleep problems, obesity, academic achievement, and emotional and behavioral problems, as well as parental stress and daytime tiredness. This study has the dual potential to expand treatment resources for young children with behavioral sleep problems and to increase our scientific understanding of the long-term consequences of early childhood sleep problems.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-71 months
* Child behavioral sleep problem, as demonstrated by a score on the Children's Sleep Habits Questionnaire (CSHQ) of at least 50, or a score of 41-49 and reported weeknight sleep of 9hrs or less per night
* English speaking parent or guardian

Exclusion Criteria:

* Sleep disordered breathing, as demonstrated by a score on the CSHQ of at least 5
* Currently taking prescribed sleep medications, psychostimulants, and/or systemic corticosteroids
* Serious medical conditions likely to affect sleep, including diabetes or cancer
* Major cognitive or developmental disorder, including autism spectrum disorder

Ages: 30 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2013-11 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in actigraphic and diary measured sleep quantity and quality measures | Baseline, 3-month follow-up
  Change in actigraphic and diary measured sleep quantity (total sleep time, nocturnal sleep time) and quality (percent wake after sleep onset) measures
Change in actigraphic and diary measured sleep quantity and quality measures | Baseline, 12-month follow-up
  Change in actigraphic and diary measured sleep quantity (total sleep time, nocturnal sleep time) and quality (percent wake after sleep onset) measures
Change in actigraphic and diary measured sleep quantity and quality measures | Baseline, 24-month follow-up
  Change in actigraphic and diary measured sleep quantity (total sleep time, nocturnal sleep time) and quality (percent wake after sleep onset) measure
Change in actigraphic and diary measured sleep quantity and quality measures | Baseline, 36-month follow-up
  Change in actigraphic and diary measured sleep quantity (total sleep time, nocturnal sleep time) and quality (percent wake after sleep onset) measures
Change in actigraphic and parent report measures of sleep onset difficulties | Baseline, 3-month follow-up
  Change in actigraphic and parent report measures of sleep onset difficulties (sleep onset latency, Child Sleep Wake Scale subscales for Going to Bed and Falling Asleep)
Change in actigraphic and parent report measures of sleep onset difficulties | Baseline, 12-month follow-up
  Change in actigraphic and parent report measures of sleep onset difficulties (sleep onset latency, Child Sleep Wake Scale subscales for Going to Bed and Falling Asleep)
Change in actigraphic and parent report measures of sleep onset difficulties | Baseline, 24-month follow-up
  Change in actigraphic and parent report measures of sleep onset difficulties (sleep onset latency, Child Sleep Wake Scale subscales for Going to Bed and Falling Asleep)
Change in actigraphic and parent report measures of sleep onset difficulties | Baseline, 36-month follow-up
  Change in actigraphic and parent report measures of sleep onset difficulties (sleep onset latency, Child Sleep Wake Scale subscales for Going to Bed and Falling Asleep)

SECONDARY OUTCOMES:
Change in child anthropometric measures | Baseline, 24-month follow-up
  Change in child anthropometric measures (BMI z-score for age and gender, waist circumference)
Change in child anthropometric measures | Baseline, 36-month follow-up
  Change in child anthropometric measures (BMI z-score for age and gender, waist circumference)
Trajectory in child anthropometric measures | Baseline, 12-month follow-up, 24-month follow-up, 36-month follow-up
  Trajectory in child anthropometric measures (BMI z-score for age and gender, waist circumference)
Change in parent-reported child behavioral and emotional symptoms and executive function | Baseline, 3-month follow-up
  Change in parent-reported child behavioral and emotional symptoms (CBCL subscores for anxious/depressed, attention, somatic complaints, and aggressive behavior) and executive function (BRIEF subscores for inhibit, shift, and emotional control)
Change in parent-reported child behavioral and emotional symptoms and executive function | Baseline, 12-month follow-up
  Change in parent-reported child behavioral and emotional symptoms (CBCL subscores for anxious/depressed, attention, somatic complaints, and aggressive behavior) and executive function (BRIEF subscores for inhibit, shift, and emotional control)
Change in parent & teacher-reported child behavioral and emotional symptoms (CBCL subscores for anxious/depressed, attention, somatic complaints, and aggressive behavior) and executive function (BRIEF subscores for inhibit, shift, and emotional control) | Baseline, 24-month follow-up
Change in parent & teacher-reported child behavioral and emotional symptoms and executive function | Baseline, 36-month follow-up
  Change in parent & teacher-reported child behavioral and emotional symptoms (CBCL subscores for anxious/depressed, attention, somatic complaints, and aggressive behavior) and executive function (BRIEF subscores for inhibit, shift, and emotional control)
Change in directly assessed performance on WJIII NU achievement battery and executive function | Baseline, 12-month follow-up
  Change in directly assessed performance on WJIII NU achievement battery (extended pre-academic battery plus oral language and basic reading skills) and executive function (iPad-based testing).
Change in directly assessed performance on WJIII NU achievement battery and executive function | Baseline, 24-month follow-up
  Change in directly assessed performance on WJIII NU achievement battery (extended pre-academic battery plus oral language, basic reading skills, math, and written expression) and executive function (iPad-based testing)
Change in directly assessed performance on WJIII NU achievement battery and executive function | Baseline, 36-month follow-up
  Change in directly assessed performance on WJIII NU achievement battery (extended pre-academic battery plus oral language, basic reading skills, math, and written expression) and executive function (iPad-based testing)
Trajectory in actigraphic and diary measured sleep quantity and quality measures | Baseline, 3-month follow-up, 12-month follow-up, 24-month follow-up, 36-month follow-up
  Trajectory in actigraphic and diary measured sleep quantity (total sleep time, nocturnal sleep time) and quality (percent wake after sleep onset) measures
Trajectory in actigraphic and parent report measures of sleep onset difficulties | Baseline, 3-month follow-up, 12-month follow-up, 24-month follow-up, 36-month follow-up
  Trajectory in actigraphic and parent report measures of sleep onset difficulties (sleep onset latency, Child Sleep Wake Scale subscales for Going to Bed and Falling Asleep)

OTHER OUTCOMES:
Change in parent-reported and actigraphic sleep hygiene behaviors | Baseline, 3-month follow-up
  Change in parent-reported and actigraphic sleep hygiene behaviors (Child Sleep Hygiene Scale total score and subscales, % of diary nights with parent in bedroom at sleep onset, mean diary-reported screen time during two hours prior to bedtime, mean actigraphic physical activity during two hours prior to bedtime, mean actigraphic light exposure during two hours prior to bedtime, mean actigraphic light exposure at nocturnal sleep midpoint)
Change in parent-reported and actigraphic sleep hygiene behaviors | Baseline, 12-month follow-up
  Change in parent-reported and actigraphic sleep hygiene behaviors (Child Sleep Hygiene Scale total score and subscales, % of diary nights with parent in bedroom at sleep onset, mean diary-reported screen time during two hours prior to bedtime, mean actigraphic physical activity during two hours prior to bedtime, mean actigraphic light exposure during two hours prior to bedtime, mean actigraphic light exposure at nocturnal sleep midpoint)
Change in survey-reported parent sleep-related beliefs and attitudes | Baseline, 3-month follow-up
  Change in survey-reported parent sleep-related beliefs and attitudes (modified MCISQ, plus outcomes expectations and self-efficacy on sleep)
Change in parent sleep and functioning via diary and survey self-report | Baseline, 3-month follow-up
  Change in parent sleep and functioning via diary and survey self-report (parent nocturnal sleep time and sleep onset latency, parent PROMIS scores for sleep disturbance, PedsQL family impact score and subscales, missed work days, productivity)
Change in parent sleep and functioning via diary and survey self-report | Baseline, 12-month follow-up
  Change in parent sleep and functioning via diary and survey self-report (parent nocturnal sleep time and sleep onset latency, parent PROMIS scores for sleep disturbance, PedsQL family impact score and subscales, missed work days, productivity)
Change in parent sleep and functioning via diary and survey self-report | Baseline,24-month follow-up
  Change in parent sleep and functioning via diary and survey self-report (parent nocturnal sleep time and sleep onset latency, parent PROMIS scores for sleep disturbance, PedsQL family impact score and subscales, missed work days, productivity)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Garrison, PhD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Research Institute, Seattle, Washington, United States